CLINICAL TRIAL: NCT02322437
Title: Home Treatment for Acute Psychiatric Care in the Canton of Aargau (Switzerland): A Randomized Controlled Trial
Brief Title: Home Treatment for Acute Psychiatric Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Psychiatric Services Aargau AG (Other)
Collaborators: Hugo & Elsa Isler Foundation (Unknown)
Responsible Party: Principal Investigator, Niklaus Stulz, PhD, Psychiatric Services Aargau AG
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PDAG-0001
Record Dates: First submitted 2014-12-11; First posted 2014-12-23 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Mental Disorders
MeSH Terms: conditions — Mental Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home treatment (Experimental): Patients in need of acute psychiatric inpatient care are treated at their houses by mobile treatment teams instead of treatment at mental hospitals whenever home treatment is possible and appropriate.
  Interventions: Other: Home treatment
- Treatment as usual (Active Comparator): Patients in need of acute psychiatric inpatient care are treated at a mental hospital.
  Interventions: Other: Treatment As Usual

INTERVENTIONS:
Other: Home treatment — Patients are treated at home whenever possible and appropriate
  Arms: Home treatment
Other: Treatment As Usual — Patients are treated at a mental hospital
  Arms: Treatment as usual

SUMMARY:
This study aims to evaluate whether psychiatric home treatment is an effective and efficient alternative to acute inpatient care in mental hospitals. A one-year prevalence cohort of psychiatric patients in need of hospitalization are randomly assigned to either treatment at inpatient wards (treatment as usual) or a new care model with the additional option of treating patients at their homes by mobile care teams. The primary focus is on checking whether optional home treatment leads to a reduction of inpatient days during a two-year follow-up period. In addition, the two service models will be compared regarding treatment cost and outcomes as well as satisfaction of patients and their relatives with psychiatric care.

Furthermore, a sub-cohort of randomly chosen patients from the prevalence-cohort will be examined by a highly trained clinical assessor to test and verify the diagnoses and the clinical ratings made by the staff members of the mental hospital under routine everyday conditions.

DETAILED DESCRIPTION:
This study aims to evaluate whether psychiatric home treatment is an effective and efficient alternative to acute inpatient care in mental hospitals. A one-year prevalence cohort of psychiatric patients in need of hospitalization are randomly assigned to either treatment at inpatient wards (treatment as usual) or a new care model with the additional option of treating patients at their homes by mobile care teams. The primary focus is on checking whether optional home treatment for crisis intervention leads to a reduction of inpatient days during a two-year follow-up period. In addition, the two service models will be compared regarding treatment cost and outcomes as well as satisfaction of patients and their relatives with psychiatric care.

Furthermore, a sub-cohort of randomly chosen patients from the prevalence-cohort will be examined by a highly trained clinical assessor to test and verify the diagnoses (SCID-I and SCID-II) and the clinical ratings (HoNOS) made by the staff members of the mental hospital under routine everyday conditions.

ELIGIBILITY:
Inclusion Criteria:

* Need for acute psychiatric inpatient care
* Residence in the canton of Aargau
* Living within 30 minutes (by car) from the headquarters of the home treatment team
* Health insurance with tarifsuisse

Exclusion Criteria:

* Insufficient proficiency in German
* Main diagnosis F0 or F1 (ICD-10)
* Patients of the forencic departement
* Patients of the child and adolescent department

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 707 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Number of inpatient days | 2 years follow-up

SECONDARY OUTCOMES:
Total days in treatment (inpatient + home treatment) | 2 years follow-up
Direct treatment costs | 2 years follow-up
Health of the Nation Outcome Scales (HoNOS) | Intake and discharge from treatment episode (expected average of 4 weeks)
  Participants will be followed for the duration of hospital stay, an expected average of 4 weeks.
Brief Symptom Checklist (BSCL) | Intake and discharge from treatment episode (expected average of 4 weeks)
  Participants will be followed for the duration of hospital stay, an expected average of 4 weeks.
Perceptions of Care-18 | Discharge from treatment episode (expected average of 4 weeks)
  Participants will be assessed at discharge from hospital, after an expected average of 4 weeks.
Satisfaction of patients' relatives | Discharge from treatment episode (expected average of 4 weeks)
  Relatives' satisfaction will be assessed with an adapted version of the Perceptions of Care-18 questionnaire at discharge of the patients from hospital, after an expected average of 4 weeks. The proportion of satisfied relatives will be reported for both study arms.
Number of rehospitalizations per patient | 2 years follow-up
Number of patients with adverse events | 2 years follow-up
  E.g. suicide or attempted suicide.

CONTACTS AND LOCATIONS:
Overall Officials: Niklaus Stulz, PhD, Principal Investigator — Psychiatric Services Aargau AG
Locations (1):
- Psychiatric Services Aargau AG, Brugg, Canton of Aargau, Switzerland

REFERENCES:
- [Derived] Stulz N, Wyder L, Maeck L, Hilpert M, Lerzer H, Zander E, Kawohl W, Grosse Holtforth M, Schnyder U, Hepp U. Home treatment for acute mental healthcare: randomised controlled trial. Br J Psychiatry. 2020 Jun;216(6):323-330. doi: 10.1192/bjp.2019.31. PMID 30864532